CLINICAL TRIAL: NCT05547581
Title: Early Detection of Contrast Induced Nephropathy After Coronary Angiography : Predictive Value of Osteopontin
Brief Title: Predictive Value of Osteopontin for Contrast Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Noura gamal (Other)
Responsible Party: Sponsor-Investigator, Noura gamal, Director,assistant lecture,principle investigator.clinical physician., Assiut University
Organization: Assiut University (Other)
Other Study IDs: CIN
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Contrast-induced Nephropathy
Keywords: CIN

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early detection of contrast induced nephropathy by using osteopontin as an early marker for prediction

DETAILED DESCRIPTION:
People who undergo coronary angiography are at risk of contrast-associated acute kidney injury (CA-AKI) .

The prevention therapy is the main approach to address CA-AKI, minimizing the volume of contrast media and intravenous hydration before and after the procedure which may not be appropriate for those with heart failure .

Given limited treatment options once CA-AKI develops and an unfavourable associated prognosis, early identification of those at risk of CA-AKI is crucial.

Also, there is studies was linking CA-AKI with a higher mortality rate and adverse future cardiovascular events, and risk for future CA-AKI events .

Mehran and colleagues described CA-AKI risk score predicting both CA-AKI and cardiovascular events after angiographic procedures.

however, studies have also investigated the role of different biomarkers in prediction of AKI like osteopontin, in 2020, a consensus statement was released regarding how best to incorporate kidney biomarkers into clinical practice.

Osteopontin is an extracellular structural protein synthesized by various cell types like osteoblasts, smooth muscle. and found in the loop of Henle and distal nephrons in normal kidneys. Recent studies have found that osteopontin has a critical role in tubulogenesis, cell apoptosis, promotion of cell regeneration. Lorenzen and colleagues found that critically ill patients with AKI have higher osteopontin concentrations than critically ill patients without AKI.

Few studies have investigated the role of osteopontin in the detection of AKI.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing coronary with or without intervention between 2022and 2024 were prospectively enrolled at the study.

Patients were referred for angiography for various acute and nonacute indications, including acute coronary syndromes, heart failure, abnormal stress tests, stable chest pain, claudication, and routine preoperative evaluation.

Patient with CKD stage 1 or 2 only

Exclusion Criteria:

* Pt has history of contrast induced nephropathy before. Patient known to have Chronic kidney disease stage 3A upto 5D Pt has contraindication for coronary angiograghy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sample size 155 at effect size 0.2 power 80 and alfa error 0.05
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2022-12-07 (Estimated); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
early detection of patients at risk of (CA-AKI) before angiographic procedures | Baseline
  Early prediction of CIN for early prevention and proper management

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sobh, Study Director — Assiut University

REFERENCES:
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Pucelikova T, Dangas G, Mehran R. Contrast-induced nephropathy. Catheter Cardiovasc Interv. 2008 Jan 1;71(1):62-72. doi: 10.1002/ccd.21207. PMID 17975790
- [Background] Ibrahim NE, McCarthy CP, Shrestha S, Lyass A, Li Y, Gaggin HK, Simon ML, Massaro JM, D'Agostino RB Sr, Garasic JM, van Kimmenade RR, Januzzi JL Jr. Blood kidney injury molecule-1 predicts short and longer term kidney outcomes in patients undergoing diagnostic coronary and/or peripheral angiography-Results from the Catheter Sampled Blood Archive in Cardiovascular Diseases (CASABLANCA) study. Am Heart J. 2019 Mar;209:36-46. doi: 10.1016/j.ahj.2018.12.001. Epub 2018 Dec 7. PMID 30641399
- [Background] Mehran R, Owen R, Chiarito M, Baber U, Sartori S, Cao D, Nicolas J, Pivato CA, Nardin M, Krishnan P, Kini A, Sharma S, Pocock S, Dangas G. A contemporary simple risk score for prediction of contrast-associated acute kidney injury after percutaneous coronary intervention: derivation and validation from an observational registry. Lancet. 2021 Nov 27;398(10315):1974-1983. doi: 10.1016/S0140-6736(21)02326-6. Epub 2021 Nov 15. PMID 34793743
- [Background] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Background] Ostermann M, Zarbock A, Goldstein S, Kashani K, Macedo E, Murugan R, Bell M, Forni L, Guzzi L, Joannidis M, Kane-Gill SL, Legrand M, Mehta R, Murray PT, Pickkers P, Plebani M, Prowle J, Ricci Z, Rimmele T, Rosner M, Shaw AD, Kellum JA, Ronco C. Recommendations on Acute Kidney Injury Biomarkers From the Acute Disease Quality Initiative Consensus Conference: A Consensus Statement. JAMA Netw Open. 2020 Oct 1;3(10):e2019209. doi: 10.1001/jamanetworkopen.2020.19209. PMID 33021646
- [Background] PubMed